CLINICAL TRIAL: NCT06186895
Title: Dexmedetomidine Versus Fentanyl on Postoperative Analgesic Profile in Patients With Morbid Obesity Undergoing Laparoscopic Sleeve Gastrectomy
Brief Title: Dexmedetomidine Versus Fentanyl on Postoperative Analgesic Profile in Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Doha Mohammed Bakr, Lecturer of anesthessiology, surgical intensive care and pain medicine, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-6-2020
Record Dates: First submitted 2023-12-17; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Pain, Postoperative
Keywords: Dexmedetomidine, fentanyl, analgesia,Sleeve Gastrectomy
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine group (Experimental): Group D, received an intravenous loading dose of DEX (1 μg/kg) over 15 minutes prior to the anesthetic induction. Following the intubation procedure, a maintenance infusion of DEX was delivered at a rate of 0.6 μg/kg/h. The infusion was discontinued upon trocars removal
  Interventions: Drug: Dexmedetomidine
- Fentanyl group (Active Comparator): Group F were administered fentanyl (1 μg/kg) that was given intravenously slowly over 60 seconds before induction of anesthesia as a loading dose. Following intubation, a continuous infusion of fentanyl was administered at a rate of 1μg/kg/hr. The infusion was discontinued upon the removal of the trocars.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — received an intravenous loading dose of DEX (1 μg/kg) over 15 minutes prior to the anesthetic induction. Following the intubation procedure, a maintenance infusion of DEX was delivered at a rate of 0.6 μg/kg/h. The infusion was discontinued upon trocars removal.
  Arms: Dexmedetomidine group
Drug: Fentanyl — fentanyl (1 μg/kg) that was given intravenously slowly over 60 seconds before induction of anesthesia as a loading dose. Following intubation, a continuous infusion of fentanyl was administered at a rate of 1μg/kg/hr. The infusion was discontinued upon the removal of the trocars.
  Arms: Fentanyl group

SUMMARY:
Dexmedetomidine (Dex) activates the α2 adrenergic receptor that is present within the locus coeruleus, leading to anxiolysis, hypnosis, analgesia, and sedation.

We conducted our research to compare the effects of fentanyl and DEX on the postoperative analgesic profile and complications in morbidly obese patients after sleeve gastrectomy.

DETAILED DESCRIPTION:
The participants were assigned to two groups of equal size (32 patients in each group) by the use of computer-generated numbers and sealed opaque envelopes. The participants allocated to the DEX group, also known as Group D, received an intravenous loading dose of DEX (1 μg/kg) over 15 minutes prior to the anesthetic induction. Following the intubation procedure, a maintenance infusion of DEX was delivered at a rate of 0.6 μg/kg/h. The infusion was discontinued upon trocars removal. The patients assigned to the fentanyl group (referred to as Group F) were administered fentanyl (1 μg/kg) that was given intravenously slowly over 60 seconds before induction of anesthesia as a loading dose. Following intubation, a continuous infusion of fentanyl was administered at a rate of 1μg/kg/hr. The infusion was discontinued upon the removal of the trocars.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) of 35 kg/m2 or more.
* American Society of Anesthesiology (ASA) physical status of II-III.
* all participants would have a laparoscopic sleeve gastrectomy (LSG).

Exclusion Criteria:

* allergy to α2 -adrenergic agonist.
* kidney, liver, neuromuscular disorders, and cardiac disease.
* or patients on opioid medications.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
visual analogue score | from arrival to PACU until 12 hours after surgery
  visual analogue pain score (VAS) from 0-10 (0: no pain, 10: the worst pain). It was assessed in post anesthesia care unit ( PACU) and every 2 hours for 12 hours postoperatively

SECONDARY OUTCOMES:
The time of the first analgesic request | first postoperative day
the total opioid dose consumed during the first 12 hours postoperatively | 12 hours after surgery
incidence of nausea and vomiting | 2 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ryad Ghoraba, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after publishing, the information will be accessible on demand
Supporting Information: Study Protocol
Time Frame: after publishing